CLINICAL TRIAL: NCT06212570
Title: KeyScope: First-In-Human Clinical Study for Cancer Diagnosis in Uganda
Brief Title: KeyScope Study in Uganda
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Makerere University (Other); Uganda Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00110170
Record Dates: First submitted 2023-11-27; First posted 2024-01-19 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Abdominal Neoplasm
MeSH Terms: conditions — Abdominal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KeySuite (Experimental): The KeyLoop and KeyScope devices will be used to perform intra-abdominal biopsies.
  Interventions: Device: KeySuite

INTERVENTIONS:
Device: KeySuite — KeyScope and KeyLoop will be used to perform biopsies of intra-abdominal masses and cancers.

SUMMARY:
KeyScope and KeyLoop (collectively called KeySuite) are laparoscopic prototypes that the investigators have designed for the resources, needs and challenges of low- and middle- income countries (LMICs). KeyScope is a laparoscope that plugs into a laptop computer to display images during surgery. It links to a telementoring application so that experienced surgeons can mentor surgeons in capacity-building partnerships. KeyLoop is a laparoscopic retractor that lifts the abdominal wall during surgery, obviating the need for a constant power supply and medical-grade carbon dioxide.

The investigators will perform a clinical First-in-Human study at the Uganda Cancer Institute. Ugandan surgeons will use the KeySuite devices to perform biopsies of intra-abdominal tumors.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of intra-abdominal mass suspicious for cancer
* body mass index (BMI) of 18-30
* weight 20-100kg
* biopsy necessary to determine cancer diagnosis and classify pathology
* surgeon determine that laproscopic biopsy it technically appropriate

Exclusion Criteria:

* significant comorbidities
* previous major abdominal surgery
* current pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Establish the clinical safety KeySuite | Day of surgery
  This will be determined by whether or not the procedure was able to be completed laproscopically or had to be converted to open surgery.

SECONDARY OUTCOMES:
Time to complete surgery | Day of surgery
  Length of surgery will be recorded
Estimated blood loss | Day of surgery
  Blood loss will be recorded
Surgical injuries and adverse events | Day of surgery
  Surgical injuries (device-related and unrelated) and other adverse events at the time of surgery will be recorded

OTHER OUTCOMES:
Surgical site infection | 30 days
  Any infections at the surgical site will be recorded and followed until resolution
Post-operative complications | 30 days
  All post-operative complications will be recorded
Mortality | 30 days
  Survival through 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Fitzgerald, MD, PhD, Principal Investigator — Duke Health
Locations (1):
- Uganda Cancer Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No